CLINICAL TRIAL: NCT03651206
Title: An International Multicentric Randomized Phase II Evaluating Dostarlimab in Combination With Niraparib Versus Niraparib Alone Compared to Chemotherapy in the Treatment of Metastatic or Recurrent Endometrial or Ovarian Carcinosarcoma After at Least One Line of Chemotherapy
Brief Title: Recurrent Ovarian CarcinoSarcoma Anti-pd-1 Niraparib
Acronym: ROCSAN
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: ARCAGY/ GINECO GROUP (Other)
Collaborators: Tesaro, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ENGOT-en8
Record Dates: First submitted 2018-08-20; First posted 2018-08-29 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Ovarian Carcinosarcoma; Endometrial Carcinosarcoma
Keywords: Malignant mixed Mullerian tumors; Metastatic ovarian carcinosarcoma; Recurrent ovarian carcinosarcoma; Metastatic endometrial carcinosarcoma; Recurrent endometrial carcinosarcoma; Niraparib; TSR-042 (Dostarlimab)
MeSH Terms: interventions — niraparib; dostarlimab; Antineoplastic Agents

STUDY DESIGN:
Intervention Model Description: Phase 2 :
  Arm A - Niraparib
  Arm B - Niraparib plus TSR-042
  Arm C - Chemotherapy drugs
  Peak the winner between the Arm A or the arm B
  Phase 3:
  Single arm - Niraparib plus TSR-042
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm A - Niraparib (Experimental): Niraparib, 200 mg or 300 mg, daily dose
  Interventions: Drug: Niraparib
- Arm B - Niraparib + TSR-042 (Dostarlimab) (Experimental): Niraparib, 200 mg or 300 mg, daily dose
  TSR042, intravenous infusion on Day 1 of every 21-day cycle at 500 mg for the 4 first cycles, followed by 1,000 mg on Day 1 of every 42-day cycle thereafter
  Interventions: Combination Product: Niraparib + TSR-042 (Dostarlimab)
- Arm C - Chemotherapy drugs (Active Comparator): Chemotherapies (Standard of care)
  For Ovarian Cancer Patients Paclitaxel, 80 mg/m², Intravenous, Day 1, 8, 15 every 28 days Pegylated Liposomal Doxorubicin, 40 mg/m², Intravenous, every 28 days Topotecan, 4mg/m², Intravenous, Day 1, 8, 15 every 28 days
  For Endometrial Cancer Patients Doxorubicin, 60 mg/m², Intravenous, every 21 days Paclitaxel, 80 mg/m², Intravenous, Day 1, 8, 15 every 28 days Gemcitabine, 800 mg/m², Intravenous, Day 1, 8 every 21 days
  Interventions: Drug: Chemotherapy Drugs

INTERVENTIONS:
Drug: Niraparib — PARP Inhibitor
  Arms: Arm A - Niraparib
Combination Product: Niraparib + TSR-042 (Dostarlimab) — Combination of 2 drugs, a PARP Inhibitor and an Anti-PD-1
  Arms: Arm B - Niraparib + TSR-042 (Dostarlimab)
Drug: Chemotherapy Drugs — Chemotherapies given in standard of care
  Arms: Arm C - Chemotherapy drugs

SUMMARY:
Carcinosarcomas (CS) (malignant mixed Müllerian tumors) are highly aggressive and rare tumors with a worldwide annual incidence between 0.5-3.3 cases/100.000 women. Gynecological CS, i.e. ovarian CS (OCS) and uterine CS (UCS), have a 5-year overall survival (OS) < 10% and a poor prognosis. After initial treatment (surgery +/- adjuvant radiotherapies +/- chemotherapies (CT)), vast majority of patients relapsed and received diverse CT producing modest benefits, and nearly all patients will die. After first line CT including platinum salt, monotherapy (doxorubicin or paclitaxel) is frequently used for relapsed patients, but the response rate (RR) is <20%, progression-free survival (PFS) <4 months, and OS <1 year. In this unmet need situation, a better knowledge of these aggressive neoplasms is essential to propose new therapeutic options.

ELIGIBILITY:
Inclusion Criteria:

1. Progressive or recurrent uterine or ovarian carcinosarcoma (Malignant Mixed Mullerian Tumor-MMMT).
2. The primary diagnosis must be histologically confirmed and central pathological review of the initial tumor or biopsy at relapse will be done.
3. Mandatory tumor samples: Availability of tumor sample(s) from a recently (not older than 3 months) obtained archival FFPE tumor tissue block or agreement for having a new tumor biopsy if lesion amenable, with ≥ 20% cellularity and tumoral surface ≥ 8 mm².
4. Progressive disease as defined by RECIST 1.1., within 12 months from last chemotherapy cycle.
5. Failure after ≥1 prior platinum containing regimen, which may have been given in the adjuvant setting.
6. Patient must have had 1 prior chemotherapeutic regimen for management of carcinosarcoma that may have included chemotherapy, chemotherapy and radiotherapy, and/or consolidation/maintenance therapy.
7. Patient must be free of active infection requiring antibiotics.
8. Any hormonal therapy directed at the malignant tumor must be discontinued at least one week prior to beginning protocol chemotherapy; continuation of hormone replacement therapy is permitted.
9. Patient must have ECOG Performance Status ≤2.
10. Life expectancy of > 2 months.
11. Adequate bone marrow function:

    * Platelet count greater than or equal to 100,000/mm3
    * Absolute neutrophil count (ANC) greater than or equal to 1,500/mm3
    * Hemoglobin > 9g/dL
12. Adequate hepatic and renal function:

    * Total bilirubin ≤1.5x Upper Limit of Normal (ULN) unless liver metastases are present, in which case they must be ≤3x ULN (≤2.0 in patients with known Gilberts syndrome OR direct bilirubin ≤ 1 x ULN)
    * Serum creatinine ≤1.5x upper limit of normal (ULN) or calculated creatinine clearance ≥ 60 mL/min using Cockcroft-Gault equation
    * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5x ULN unless liver metastases are present, in which case they must be ≤5x ULN
    * Alkaline phosphatase < 2.5 times ULN
    * Serum albumin > 3 g/dL
13. International normalized ratio (INR) or prothrombin time (PT) ≤1.5× ULN unless patient is receiving anticoagulant therapy as long as PT or partial thromboplastin (PTT) is within therapeutic range of intended use of anticoagulants. Activated partial thromboplastin time (aPTT) ≤1.5× ULN unless patient is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants.
14. Patient must have normal BP or adequately treated and controlled hypertension (systolic BP≤140 mmHg and/or diastolic BP ≤90 mmHg)
15. Patient receiving corticosteroids may continue as long as their dose is stable and ≤10mg/day (prednisone equivalent) for at least 4 weeks prior to initiating protocol therapy.
16. Patient must agree to not donate blood during the study or for 90 days after the last dose of study treatment.
17. Left ventricular ejection fraction (LVEF) > Lower Limit of Normal (LLN) as assessed by either multigated acquisition (MUGA) scan or echocardiogram (ECHO), for patients planned to receive Anthracycline based therapy.
18. 18. Patient has a negative urine or serum pregnancy test within 7 days prior to taking study treatment if of childbearing potential and agrees to abstain from activities that could result in pregnancy from screening through 180 days after the last dose of study treatment, or is of nonchildbearing potential.

    * Non-childbearing potential is defined as follows:

      * ≥45 years of age and has not had menses for >1 year
      * Patients who have been amenorrhoeic for <2 years without history of a hysterectomy and oophorectomy must have a follicle stimulating hormone value in the postmenopausal range upon screening evaluation
      * Post-hysterectomy, post-bilateral oophorectomy, or post-tubal ligation. Documented hysterectomy or oophorectomy must be confirmed with medical records of the actual procedure or confirmed by an ultrasound. Tubal ligation must be confirmed with medical records of the actual procedure.
    * For women of childbearing potential: the patient must be willing to use a highly effective contraception measure throughout the study, starting with the screening visit through 180 days after the last dose of study treatment. See Section 4.3. for a list of highly effective contraception methods. Information must be captured appropriately within the site's source documents. Note: Abstinence is acceptable if this is the established and preferred contraception for the patient.
19. Patient must agree to not breastfeed during the study and for 180 days after the last dose of study treatment.
20. Patient able to take oral medications.
21. 21. Female aged ≥18 years at time of signing ICF.
22. Patient must have signed an approved informed consent.
23. For France only: patient affiliated to, or a beneficiary of, a social security category.

Exclusion Criteria:

1. Not enrolled in any interventional clinical trial (except to biological trials that must be validated by the sponsor).
2. Prior treatment with niraparib or other PARPi therapy or PD1/PDL-1 inhibitors.
3. Patient has had investigational therapy, immunotherapy, chemotherapy or biological therapy administered within 4 weeks or within a time interval less than at least 5 half-lives of the investigational agent, whichever is longer, prior to randomization. Patient has had radiotherapy within 4 weeks prior to randomization.
4. Patient must not have had major surgery ≤ 3 weeks prior to initiating protocol therapy and participant must have recovered from any surgical effect.
5. Previous treatment with the chemotherapy regimen selected as the control arm by the investigator.

   * Prior therapy with paclitaxel given on a three-weekly regimen is permitted for patients receiving weekly Paclitaxel.
   * Prior treatment with weekly paclitaxel is permitted where this has been used as part of first line therapy and it is greater than 6 months since the last dose of weekly paclitaxel.
   * Prior weekly paclitaxel for relapsed disease is not permitted.
6. Patients who have received more than 3 prior cytotoxic chemotherapies for management of uterine or ovarian carcinosarcoma.
7. Patients with persistent, clinically significant > Grade 1 toxicity.
8. Patient has clinically significant cardiovascular disease (eg, significant cardiac conduction abnormalities, uncontrolled hypertension, myocardial infarction, uncontrolled cardiac arrhythmia or unstable angina < 6 months to enrollment, NHYA grade 2 or greater congestive heart failure, serious cardiac arrhythmia requiring medication, Grade 2 or greater peripheral vascular disease, and history of cerebrovascular accident within 6 months)
9. Patients with any other severe concurrent disease, which may increase the risk associated with study participation or study drug administration and, in the judgment of the investigator, would make the patient inappropriate for entry into this study, including significant neurologic, psychiatric, infectious, hepatic, renal, or gastrointestinal diseases or laboratory abnormality. Examples include, but are not limited to, uncontrolled ventricular arrhythmia, recent (within 90 days) myocardial infarction, uncontrolled major seizure disorder, unstable spinal cord compression, superior vena cava syndrome, or any psychiatric disorder that prohibits obtaining informed consent.
10. Symptoms or signs of gastrointestinal obstruction requiring parenteral nutrition or hydration or any other gastro-intestinal disorders or abnormalities, including difficulty swallowing, that would interfere with drug absorption.
11. Patient experienced ≥ Grade 3 immune-related AE with prior immunotherapy, with the exception of non-clinically significant lab abnormalities
12. Participant has had radiation therapy encompassing >20% of the bone marrow within 2 weeks prior to Day 1 of protocol therapy, or any radiation therapy within 1 week prior to Day 1 of protocol therapy.
13. Patient has a diagnosis of immunodeficiency or has received systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to initiating protocol therapy
14. Patient has a known history of human immunodeficiency virus (type 1 or 2 antibodies).
15. Patient has known active hepatitis B (e.g., hepatitis B surface antigen [HBsAg] reactive) or hepatitis C (e.g., hepatitis C virus [HCV] ribonucleic acid [qualitative] is detected).
16. Patient has an active autoimmune disease that has required systemic treatment in the past 2 years (ie, with use of disease-modifying agents, corticosteroids, or immunosuppressive drugs). Replacement therapy (eg, thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
17. Patient must not have a history of interstitial lung disease.
18. Patient has received a live vaccine within 14 days of initiating protocol therapy.
19. Patient must not have received a transfusion (platelets or red blood cells) ≤ 4 weeks prior to initiating protocol therapy.
20. Patient must not have received colony stimulating factors (eg, granulocyte colony-stimulating factor, granulocyte macrophage colony stimulating factor, or recombinant erythropoietin) within 4 weeks prior initiating protocol therapy.
21. Patient has had any known Grade 3 or 4 anemia, neutropenia or thrombocytopenia due to prior chemotherapy that persisted > 4 weeks and was related to the most recent treatment.
22. Patient must not have any known history of myelodysplastic syndrome (MDS) or acute myeloid leukemia (AML)
23. Symptomatic CNS metastasis or leptomeningeal carcinomatosis.
24. Patients with a history of other invasive malignancies (any evidence of other malignancy being present within the last 3 years) or with a concomitant invasive malignancy, with the exception of non-melanoma skin cancer; patients are also ineligible if their previous cancer treatment contraindicates this protocol therapy.
25. Known, hypersensitivity reactions or allergy to investigational drugs or their excipients that contraindicates the subject's participation.
26. Any psychological, familial, sociological or geographical consideration potentially hampering compliance with the study protocol and follow up schedule; those considerations should be discussed with the patient before registration in the trial.
27. Patients under psychiatric care and patients admitted to a health or social institution.
28. Patients deprived of their liberty by judicial or administrative decision.
29. Patients under a legal protection measure or unable to express their consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2020-07-15 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Response Rate (RR) at 4 months | 4 months after the last patient included
  RR is defined as the proportion of patients with a partial response or complete response 4 months after randomization
Overall survival (OS) | 1 year after the last patient included
  OS is the time from the date of the randomization until death due to any cause

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | 1 year after the last patient included
  PFS is the time from randomization to the date of event defined as the first documented progression (RECIST 1.1) or death due to any cause.
Time To Subsequent Treatment (TTST) | 1 year after the last patient included
  TTST is the time from the date of randomization to the earliest date of anti-cancer therapy start following study treatment discontinuation, or death by any cause in the absence of start of new anti-cancer therapy
Progression-Free Survival 2 (PFS2) | 1 year after the last patient included
  PFS2 is the time from the date of randomization to the second objective disease progression, or death from any cause, whichever occurs first.
Objective Response Rate (ORR) | 1 year after the last patient included
  ORR is the proportion of patients with a best response of Complete Response or Partial Response.
Adverse events | 1 year after the last patient included
  Assessed by CTCAE 5.0
Patient-reported outcomes (PROs) | 1 year after the last patient included
  Assessed with questionnaires to be completed by patient and collected frequently during the study

CONTACTS AND LOCATIONS:
Locations (36):
- France (24):
  - ICO Paul Papin, Angers
  - CHRU Jean Minjoz, Besançon
  - Centre Régional de Lutte contre le cancer - Institut Bergonié, Bordeaux
  - CHU de BREST - Hôpital Cavale Blanche, Brest
  - Centre François Baclesse, Caen
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre Georges François Leclerc, Dijon
  - Centre Oscar Lambret, Lille
  - CHU de Limoges - Hôpital Dupuytren, Limoges
  - Centre Léon Bérard, Lyon
  - Institut Paoli Calmettes, Marseille
  - Hôpital Privé du Confluent S.A.S., Nantes
  - Centre Hospitalier Universitaire de Nîmes, Institut de Cancérologie du GARD, Nîmes
  - Groupe Hospitalier des Diaconesses Croix Saint-Simon, Paris
  - Institut Curie, Paris
  - Hopital Milétrie - Centre Hospitalier Universitaire Poitiers, Poitiers
  - Centre Eugène Marquis, Rennes
  - ICO - Centre René Gauducheau, Saint-Herblain
  - CHU Saint-Etienne - Pôle de Cancérologie, Saint-Priest-en-Jarez
  - ICANS, Strasbourg
  - Hôpitaux Universitaires de Strasbourg, Strasbourg
  - IUCT Oncopole - Institut Claudius Régaud, Toulouse
  - ICL - Centre Alexis Vautrin, Vandœuvre-lès-Nancy
  - Institut Gustave Roussy, Villejuif
- Italy (8):
  - Azienda Ospedaliero-Universitaria di Bologna IRCCS Istituto di Ricerca e di Cura a Carattere Scientifico, Bologna
  - Azienda Ospedaliera Per L'Emergenza Cannizzaro, Catania
  - Istituto Romagnolo Per Lo Studio Dei Tumori Dino Amadori IRST S.r.l., Meldola
  - Ospedale San Raffaele S.r.l., Milan
  - Humanitas Mirasole S.p.A., Milan
  - IRCCS Istituto Nazionale Tumori Fondazione Pascale, Napoli
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma
  - Azienda Ospedaliera Ordine Mauriziano Di Torino, Torino
- Spain (4):
  - Hospital Universitario Ramon Y Cajal, Madrid
  - Hospital Universitario 12 De Octubre, Madrid
  - Hospital Virgen de la Arrixaca, Murcia
  - Hospital Clinico Universitario De Valencia, Valencia

IPD SHARING:
Plan to Share IPD: No
No sharing plan